CLINICAL TRIAL: NCT03999944
Title: Non-Inferiority Study of the FRESCA Airbox Positive Airway Pressure System Versus the (Predicate) FRESCA Positive Airway Pressure System for the Treatment of Obstructive Sleep Apnea
Brief Title: Non-Inferiority Study of the FRESCA Airbox Positive Airway Pressure System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FRESCA Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18-01
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, randomized crossover assignment, multi-center study conducted in the United States
Who Masked: Outcomes Assessor
Masking Description: Central sleep study scorer will be masked to assignment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sequence 1 (Other): FRESCA Airbox Flow Generator set to fixed pressure first, then FRESCA Airbox Generator set to auto-adjusting pressure.
  Second intervention within 1 - 10 days of first intervention.
  Interventions: Device: positive airway pressure system
- Sequence 2 (Other): FRESCA Airbox Flow Generator set to auto-adjusting pressure first, then FRESCA Airbox Generator set to fixed pressure.
  Second intervention within 1 - 10 days of first intervention.
  Interventions: Device: positive airway pressure system

INTERVENTIONS:
Device: positive airway pressure system — Positive Airway Pressure System

SUMMARY:
Prospective, open-label, randomized crossover assignment, multi-center non-inferiority study conducted in the United States

DETAILED DESCRIPTION:
This study is designed to demonstrate that the FRESCA Airbox Positive Airway Pressure System is non-inferior to the existing FRESCA Positive Airway Pressure System. Subjects meeting the inclusion and exclusion criteria will be randomized to one sleep night with the existing FRESCA device programmed to fixed pressure and one sleep night with the investigational FRESCA device programmed to auto-adjusting pressure and exhale pressure relief.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 22 - 75 years old.
2. BMI: ≤ 40 kg/m2.
3. Subjects diagnosed with OSA (either newly diagnosed (naive) OSA subjects or current CPAP subjects).
4. Must be able to be fitted properly with FRESCA mask.
5. Must be able to comply with all study requirements as outlined in the protocol.
6. Subject must complete a valid PSG titration night.

Exclusion Criteria:

1. Subjects with non-OSA sleep disorders (including periodic limb movement (PLM) disorder and chronic insomnia).
2. Subjects with substantial central or mixed apneas (central and mixed apnea ≥ 5/hr.).
3. Subjects with prior surgical intervention for OSA.
4. Subjects with frequent or sustained episodes of O2 saturation ≤75%.
5. Subjects with obesity-related hypoventilation.
6. Subjects currently using a CPAP full face mask.
7. Subjects who are medically unstable.
8. Subjects with unstable or severe cardiovascular abnormalities (e.g., heart failure, valvular heart disease).
9. Subjects with atrial fibrillation or other arrhythmias that are not effectively controlled with medication.
10. Subjects with hypotension or uncontrolled HTN.
11. Subjects with chronic lung disease, including COPD.
12. Subjects with significant cardiopulmonary disease.
13. Subjects with ongoing severe nasal allergies or sinusitis or difficulty breathing through the nose; persistent blockage of one or both nostrils; or any nasal or facial abnormalities that would not allow adequate placement and use of the mask.
14. Subjects with surgery of the upper airway, nose, sinus or middle ear within the previous year.
15. Subjects currently working nights, rotating night shifts or with planned travel during the study period.
16. Subjects on a non-stable dose of medications or other agents that may affect sleep and/or PSG (e.g., sedatives or hypnotics).
17. Subjects who consume > 500 mg caffeine per day (e.g., > 8 cola-type beverages, > 5 cups of coffee).
18. Subjects who consume > 14 alcoholic drinks/week.
19. Subjects who are pregnant (confirmed verbally).
20. Subjects currently enrolled in any other research study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Goetting, MD, Principal Investigator — Bronson Sleep Health
Locations (6):
- United States (6):
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - NeuroTrials Research, Atlanta, Georgia
  - Neurological Center of North GA, Gainesville, Georgia
  - Bronson Sleep Health, Portage, Michigan
  - Clinilabs Drug Development Corp, New York, New York
  - Bogan Sleep Consultants, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 subjects were screened for eligibility
Pre-assignment Details: 52 subjects were enrolled and randomized.
Groups:
- Sequence 1 (FRESCA Flow Generator Then FRESCA Airbox Flow Generator): Subject first used FRESCA Flow Generator during in-lab sleep night, then used the FRESCA Airbox Flow Generator during in-lab sleep night between 0 - 14 days later.
- Sequence 2 (FRESCA Airbox Flow Generator, Then FRESCA Flow Generator): Subject first used FRESCA Airbox Flow Generator during in-lab sleep night, then used the FRESCA Flow Generator during in-lab sleep night between 0 - 14 days later.
Period: First Sleep Night
Arm/Group | Sequence 1 (FRESCA Flow Generator Then FRESCA Airbox Flow Generator) | Sequence 2 (FRESCA Airbox Flow Generator, Then FRESCA Flow Generator)
Started | 26 | 26
Completed | 22 | 24
Not Completed | 4 | 2
Period: Second Sleep Night
Arm/Group | Sequence 1 (FRESCA Flow Generator Then FRESCA Airbox Flow Generator) | Sequence 2 (FRESCA Airbox Flow Generator, Then FRESCA Flow Generator)
Started | 22 | 24
Completed | 22 | 20
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: in] | 67.70 (3.729)
Weight [Mean (Standard Deviation); unit: lbs] | 213.98 (36.833)
BMI [Mean (Standard Deviation); unit: kg/m2] | 32.69 (4.195)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 123.26 (13.740)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 75.74 (8.267)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 72.74 (11.133)
Oral Temperature [Mean (Standard Deviation); unit: degrees F] | 97.87 (0.513)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index (AHI)
Description: The mean combined number of apnea and hypopnea events per hour of sleep
Time Frame: 1 sleep night
Population: All participants who completed two valid sleep nights were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: events/hr
Groups:
- FRESCA Flow Generator: Participants used the FRESCA Flow Generator on either the first or second sleep night.
- FRESCA Airbox Flow Generator: Participants used the FRESCA Airbox Flow Generator on either the first or second sleep night.
Arm/Group | FRESCA Flow Generator | FRESCA Airbox Flow Generator
Number analyzed (Participants) | 42 | 42
events/hr | 3.20 (8.620) | 4.86 (10.047)

2. Secondary Outcome: Oxygen Desaturation Index (ODI)
Description: The number of oxygen desaturations ≥ 4% per hour of sleep
Time Frame: 1 sleep night
Population: All participants who completed two valid sleep nights were included in the efficacy analysis
Measure: Mean (Standard Deviation); unit: events/hr
Groups:
- FRESCA Airbox Flow Generator: Participants used the FRESCA Flow Generator on either the first or second sleep night.
Arm/Group | FRESCA Flow Generator | FRESCA Airbox Flow Generator
Number analyzed (Participants) | 42 | 42
events/hr | 3.12 (9.274) | 4.69 (10.425)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: 52 intent to treat subjects were included in the safety analysis.
Groups:
- FRESCA Flow Generator: Existing FRESCA device programmed to deliver fixed pressure.
  positive airway pressure system: Positive Airway Pressure System
- FRESCA Airbox Flow Generator: Investigational FRESCA device programmed to deliver auto-adjusting pressure
  positive airway pressure system: Positive Airway Pressure System
Arm/Group | FRESCA Flow Generator | FRESCA Airbox Flow Generator
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 4/52 | 6/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FRESCA Flow Generator (N=52) | FRESCA Airbox Flow Generator (N=52)
difficulty breathing (General disorders) | 2 (2) | 3 (3)
skin/nose irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
difficulty sleeping (General disorders) | 0 (0) | 1 (1)
discomfort from headgear (General disorders) | 0 (0) | 1 (1)
dreaming of suffocating (Psychiatric disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
increased effort with inhalation and exhalation (General disorders) | 1 (1) | 1 (1)
intermittent pain to nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT03999944/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03999944/SAP_001.pdf